CLINICAL TRIAL: NCT04424654
Title: Prospective Biomarker Analysis of Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC) Undergoing Bipolar Androgen Therapy (BAT)
Brief Title: Biomarker Analysis of Castration-resistant Prostate Cancer Undergoing Bipolar Androgen Therapy
Acronym: PSMA-BAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSL-1820
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Castration-resistant prostate cancer; Bipolar androgen therapy; PSMA-PET
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone 17 beta-cypionate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bipolar Androgen Therapy (BAT) (Experimental): Testosterone cypionate 400 mg IM every 28 days for 3 cycles
  Interventions: Drug: Testosterone cypionate

INTERVENTIONS:
Drug: Testosterone cypionate — Testosterone cypionate 400 mg IM
  Other Names: Testosterone

SUMMARY:
This is an open label phase II, single-arm, biomarker multi-institutional pilot study. Men with progressive metastatic castration-resistant prostate cancer (mCRPC) who have been treated with androgen deprivation therapy (ADT) and at least one prior second generation AR-targeted therapy (either abiraterone or enzalutamide) will be enrolled in this study. All patients will receive treatment with testosterone cypionate 400 mg, intramuscular, every 28 days for a maximum of 3 cycles or limiting toxicity, if it occurs before the end of the scheduled therapy. After 3 cycles of BAT (12 weeks), patients may continue receiving this therapy off study at the discretion of the treating physician, if clinical/radiographic benefit.

During the study period, patients will have plasma collected for cell-free tumor DNA analysis and CTC ARV7 status and also will perform 68Gallium-PSMA PET at baseline and then every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed informed consent.
* Males aged 18 years of age and above.
* Histological or cytologic proof of adenocarcinoma of the prostate.
* Known castration-resistant disease, defined according to PCWG3 criteria as: castrate serum testosterone level ≤ 50 ng/dL (≤ 1.7 nmol/L). Subjects who have failed initial hormonal therapy, either by orchiectomy or by using a GnRH agonist in combination with an anti-androgen, must first progress through anti-androgen withdrawal prior to being eligible. The minimum timeframe to document failure of anti-androgen withdrawal will be 4 weeks.
* Disease progression: serum PSA progression defined as 2 consecutive increases in PSA over a previous reference value within 6 months, each measurement at least 1 week apart, or documented bone lesions by the appearance of ≥ 2 new lesions by bone scintigraphy or dimensionally measurable soft tissue metastatic lesion assessed by CT or MRI.
* Absolute PSA ≥ 1.0 ng/mL at screening.
* Must have PSA and/or radiographic progression on AT LEAST ONE novel AR- targeted therapy (abiraterone acetate, enzalutamide, apalutamide or darolutamide). One prior chemotherapy agent for mCRPC will be allowed but is not required for inclusion.
* Prior treatment with abiraterone, enzalutamide, apalutamide, darolutamide, bicalutamide, and/or ketoconazole is allowed. There is no limit on the maximum number or types of prior hormonal therapies received.
* Must be maintained on a GnRH analogue or have undergone orchiectomy.
* Radiographic evidence of metastatic disease by CT scan and/or bone scan, performed within the prior 6 months
* Karnofsky Performance Status (KPS): ≥ 80% within 14 days before start of study treatment (ECOG < 2)
* Asymptomatic or minimally symptomatic mCRPC according to Brief Pain Inventory - Short Form (BPI-SF) performed during screening: asymptomatic is defined as BPI-SF item #3 score of 0 to 1; minimally symptomatic is defined as BPI-SF item #3 score of 2 to 4.
* Archived tumor tissue obtained prior to enrollment from a metastatic tumor lesion or from a primary tumor lesion (formalin fixed paraffin-embedded [FFPE] block or unstained tumor tissue sections). Tumor sample may be from core biopsy, punch biopsy, excisional biopsy, or surgical specimen).
* Participants must have adequate organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Hemoglobin ≥ 9.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Total bilirubin within institutional upper limit of normal (ULN) (In patients with Gilbert's syndrome, total bilirubin < 1.5x institutional ULN will be acceptable)
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) within institutional upper limit of normal
  * Participants must have Creatinine Clearance estimated using the Modified Cockcroft-Gault equation of ≥ 40 mL/min: Estimated Creatinine Clearance = (140-age [years]) x weight (kg) serum creatinine (mg/dL) x 72
* Participants must have a life expectancy ≥ 6 months.
* Male participants and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination, throughout the period of taking study treatment and for 6 months after the last dose of BAT, to prevent pregnancy in a partner.
* No evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin).

Exclusion Criteria:

* External-beam radiotherapy within the last 4 weeks prior to start of study treatment.
* Prior oral anti-androgen (e.g. bicalutamide, nilutamide, enzalutamide, apalutamide, darolutamide), or androgen synthesis inhibitor (e.g. abiraterone, orteronel) within the past 4 weeks is not permitted. 5-alpha reductase inhibitor therapies are not allowed as well.
* Prior treatment with chemotherapy for the treatment of metastatic hormone- sensitive prostate cancer is allowed if the last dose of chemotherapy was ≥ 6 months prior to enrollment. In addition, one prior chemotherapy agent for mCRPC will be allowed after a minimum wash-out period of 4 weeks prior to enrollment.
* Patients who have received prior treatment with bipolar androgen therapy (e.g. testosterone, BAT).
* Pain due to metastatic prostate cancer requiring opioid therapy.
* Patients with an intact prostate AND urinary obstructive symptoms are excluded (which includes patients with urinary symptoms from benign prostatic hyperplasia (BPH).
* Patients receiving anticoagulation therapy are not eligible for study.
* Patients with prior history of an arteriovenous thromboembolic event that occurred within the last 12 months are excluded.
* Participation in another clinical study with an investigational product during the last 4 weeks.
* Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, severe and extensive spinal metastases with concern over spinal cord compression, extensive liver metastases).
* Concurrent use of other anticancer agents or treatments, with the following exceptions:
* Ongoing treatment with LHRH agonists or antagonists, denosumab or bisphosphonate (e.g. zoledronic acid) is allowed. Ongoing treatment should be kept at a stable schedule; however, if medically required, a change of dose, compound, or both is allowed.
* Any treatment modalities involving major surgery within 4 weeks prior to the start of study treatment.
* Symptomatic nodal disease, i.e. scrotal, penile or leg edema (CTCAE ≥ Grade 3).
* Patients are excluded if they have active, known brain metastases or leptomeningeal metastases.
* Patients should be excluded if they have an active, known or suspected autoimmune disease (e.g. inflammatory bowel disease, rheumatoid arthritis, autoimmune hepatitis, lupus, celiac disease). Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg/day prednisone equivalents are permitted in the absence of active autoimmune disease.
* Permitted therapies include topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g. contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed- type hypersensitivity reaction caused by contact allergen) is permitted.
* History of allergy to study drug components.
* Other primary tumor (other than CRPC) including hematological malignancy present within the last 5 years (except non-melanoma skin cancer, low-grade superficial bladder cancer, or cancers that can be cured with local treatment alone).
* Has imminent or established spinal cord compression based on clinical findings and/or MRI.
* Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous, including, but not limited to:

  * Any uncontrolled major infection.
  * Cardiac failure NYHA (New York Heart Association) III or IV.
* Persistent toxicities (CTCAE > Grade 2) caused by previous cancer therapy, excluding alopecia.
* Poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 12 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease, or any psychiatric disorder that prohibits obtaining informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Ga68-PSMA uptake and response to Bipolar Androgen Therapy (BAT) | 12 weeks
  To evaluate the correlation between baseline Galium68-PSMA/PET maximal standard uptake value (SUVmax) and response to bipolar androgen therapy based on Prostate Cancer Working Group 3 (PCWG3).

SECONDARY OUTCOMES:
PSMA SUV kinetics during BAT | 12 weeks
  To describe the median Galium68-PSMA/PET SUVmax value variation after bipolar androgen therapy
ARV7 status and response to BAT | 12 weeks
  To evaluate the correlation between the AR-V7 status and response to bipolar androgen therapy based on Prostate Cancer Working Group 3 (PCWG3).
AR mutational status and response to BAT | 12 weeks
  To evaluate the correlation between the presence of AR mutations and response to bipolar androgen therapy based on Prostate Cancer Working Group 3 (PCWG3).
ARV7 status kinetics during BAT | 12 weeks
  To describe the ARV7 conversion rate from positive to negative after bipolar androgen therapy.
cfDNA kinetics during BAT | 12 weeks
  To describe the median cfDNA value variation after bipolar androgen therapy
Quality of life of patients receiving BAT (BPI-SF) | 12 weeks
  To evaluate quality of life using the BPI-SF questionnaire before and after BAT.
Quality of life of patients receiving BAT (EQ-5D-3L) | 12 weeks
  To evaluate quality of life using the EQ-5D-3L questionnaire before and after BAT.
Quality of life of patients receiving BAT (FACT-P) | 12 weeks
  To evaluate quality of life using the FACT-P questionnaire before and after BAT.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Sirio-Libanes, São Paulo

REFERENCES:
- [Derived] Gongora ABL, Marshall CH, Velho PI, Lopes CDH, Marin JF, Camargo AA, Bastos DA, Antonarakis ES. Extreme Responses to a Combination of DNA-Damaging Therapy and Immunotherapy in CDK12-Altered Metastatic Castration-Resistant Prostate Cancer: A Potential Therapeutic Vulnerability. Clin Genitourin Cancer. 2022 Apr;20(2):183-188. doi: 10.1016/j.clgc.2021.11.015. Epub 2021 Dec 24. No abstract available. PMID 35027313